CLINICAL TRIAL: NCT01388062
Title: e- Ab Sensor - Based Real-time Diagnosis of Influenza Virus
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Double | Purpose: Diagnostic
Other Study IDs: 201007054R
Record Dates: First submitted 2011-07-01; First posted 2011-07-06 (Estimated); Last update posted 2012-12-27 (Estimated); Status verified 2012-11

CONDITIONS: Influenza Caused by Unspecified Influenza Virus
Keywords: influenza virus

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- virus detection (Experimental)
  Interventions: Device: Electrosensing antibody probing system (e- Ab sensor)

INTERVENTIONS:
Device: Electrosensing antibody probing system (e- Ab sensor) — Electrosensing antibody probing system (e- Ab sensor), which was developed for the rapid and sensitive detection of hapten, proteins, or viral antigen in medical samples, will be used for analyzing the interaction kinetics between anti- influenza virus antibody and its antigen (influenza virus) present in patients. The system incorporates the use of engineered semiconductive antibodies or virus in vertical and lateral chip (eAbchip) or lateral flow through (eAbsignal) formats. In electrosensing antibody probing, semiconductive antibodies are bound as a suitable electrosensing probe, which specifically and selectively binds targeted molecules (influenza virus) in the test specimens. From assessment of the electric signature of semiconductive anti- influenza virus antibodies, the eABprobe could offer sensitive detection and precise quantification of EV71.

SUMMARY:
The purpose of this study is to develop a real-time diagnostic technique with e- Ab sensor for influenza virus detection, the investigators conduct a prospective clinical study. In comparison with results from direct sequencing of influenza virus, the investigators evaluate the performance of e- Ab sensor, including reproducibility, sensitivity, specificity, and cross-reaction. The potential factors which may interfere with the results would be investigated. With such technique, the investigators hope to make early diagnosis and give influenza virus patients early treatment to reduce the complications and case-fatality rate.

DETAILED DESCRIPTION:
Since April 15 and 17, 2009, when the first two cases of novel influenza A (H1N1) infection were identified in two southern California counties, as of 12 March 2010, the virus has spread to more than 213 countries and overseas territories or communities where it has caused the deaths of at least 16713 people. Therefore, a rapid diagnosis is clinically necessary and can provide clinicians the rapid answers and make early treatment possible to reduce the complications and case-fatality rate. In addition, early diagnosis of the patients will alert parents and public health workers to prevent the contacts earlier and to limit the influenza spread.

Electrosensing antibody probing system (e- Ab sensing), which was developed for the rapid and sensitive detection of hapten, proteins or viral antigen in medical samples, will be used for analyzing the interaction kinetics between Q.anti-influenza-virus and its influenza virus antigen present in flu patients'and normal samples. The system incorporates the use of engineered semiconductive antibodies or virus in vertical and lateral chip (eVchip) or lateral flow through (eVsignal) formats. In electrosensing antibody probing, semiconductive antibodies are bound as a suitable electrosensing probe which specifically and selectively binds influenza-virus epitope target molecules in the test samples.

The investigators evaluate the performance of e- Ab sensor, including reproducibility, sensitivity, specificity, and cross-reaction. The potential factors which may interfere with the results would be investigated. e- Ab sensor threshold decisions must maximize its sensitivity. Therefore, the threshold value in the test group is to find the decision could have 90% sensitivity and 90% specificity. With such technique, the investigators hope to make early diagnosis and give influenza patients early treatment to reduce the complications and case-fatality rate.

ELIGIBILITY:
Inclusion Criteria:

* A: The patients with confirmed or suspected infection.
* B: The patients without disease.

Exclusion Criteria:

* Patients will be excluded if they couldn't sign the consent.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2010-08; Primary Completion 2013-07 (Estimated); Study Completion 2013-10 (Estimated)

PRIMARY OUTCOMES:
The performance of e- Ab sensor | 1 Day
  In comparison with results from direct sequencing of influenza virus, we evaluate the performance of e- Ab sensor, including reproducibility, sensitivity, specificity, and cross-reaction.

CONTACTS AND LOCATIONS:
Overall Officials: Luan-Yin Chang, MD,PhD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan